CLINICAL TRIAL: NCT07057037
Title: Multi-center, Single Arm, Unenhanced MRI-controlled Phase III Study for Efficacy and Safety of MR Arthrography Using the NEMO-103 Injection in Patients With Known or Suspected Shoulder Joint Diseases Requiring MR Arthrography
Brief Title: Phase 3 Study of the Efficacy and Safety of MR Arthrography Using the NEMO-103 Injection in Patients With Known or Suspected Shoulder Joint Diseases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inventera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVT-NEM_P3_24
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tear; Labral Tear; Rotator Cuff Tendinosis; Rotator Cuff Tendonitis; Articular Cartilage Injury; Glenohumeral Ligament; Long Head Biceps Tendon Tear; Adhesive Capsulitis
Keywords: contrast agent; contrast enhancement in magnetic resonance imaging; Magnetic Resonance Arthrography
MeSH Terms: conditions — Rotator Cuff Injuries; Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEMO-103 Injection (Experimental)
  Interventions: Drug: NEMO-103 Injection

INTERVENTIONS:
Drug: NEMO-103 Injection — 15mL(at least 12mL), solution for Intravenous injection, single dose

SUMMARY:
The goal of this Phase 3 clinical trial is to evaluate whether MR arthrography enhanced with NEMO-103 injection (NEMO-103 Inj.) provides superior diagnostic imaging quality compared to unenhanced MRI in patients with known or suspected shoulder joint disorders, such as rotator cuff tendon tears, labral tears, and articular cartilage injuries.

⦁ The primary objective is to determine whether NEMO-103 Inj.-enhanced MR arthrography offers improved imaging quality in terms of joint distension, contrast resolution, and image sharpness compared to standard unenhanced MRI.

Participation Details:

* Each participant will undergo two MRI scans: one unenhanced and one enhanced with NEMO-103 Inj.
* NEMO-103 Inj. will be administered once, during the second study visit.
* Participants will attend a total of three site visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years at the time of informed consent.
2. Suspected or known shoulder joint diseases requiring MRA for diagnosis or evaluation at screening.
3. Voluntarily decided to participate in the study and provided written consent after receiving a sufficient explanation about this study and after fully understanding the information.

Exclusion Criteria:

1. Subjects with contraindications to MRI
2. Subjects expected to be clinically unstable during the study
3. Subjects who have received or used another IP or investigational device within 4 weeks or ≥5 half-lives, whichever is longer, prior to informed consent.
4. Pregnant or breast-feeding women, or women of childbearing potential and men who do not agree to use appropriate methods of contraception during the study.
5. Determined to be ineligible to participate in the study by the investigator due to any other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Qualitative Image Quality Metrics (Distension, Contrast, Sharpness) to Be Evaluated by Independent Central Readers | 1day procedure
  The qualitative image quality metrics (distension, contrast, and sharpness) will be assessed on a 3-point scale (good, fair, poor) for both unenhanced MRI and NEMO-103 Inj.-enhanced MR arthrography. These metrics will evaluate the degree of joint distension, the sharpness of joint margins, and the contrast between joint fluid and surrounding structures.

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System, Severance Hospital, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi